CLINICAL TRIAL: NCT00690768
Title: Pars Plana Vitrectomy (PPV) Versus Preoperative Intravitreal Bevacizumab Plus PPV for Diabetic Tractional Retinal Detachment (IBETRA Study)
Brief Title: Pars Plana Vitrectomy (PPV) Versus Preoperative Intravitreal Bevacizumab Plus PPV to Treat Diabetic Tractional Retinal Detachment (IBETRA)
Acronym: IBETRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBETRA
Record Dates: First submitted 2008-05-30; First posted 2008-06-05 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Retinopathy; Retinal Detachment
Keywords: Diabetic Retinopathy; Retinal detachment; Vitreous Hemorrhage; Bevacizumab; preoperative; pars plana vitrectomy
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Detachment; Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Preoperative Intravitreal bevacizumab and pars plana vitrectomy
  Interventions: Drug: Bevacizumab; Procedure: pars plana vitrectomy
- B (Active Comparator): Pars plana vitrectomy only
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Drug: Bevacizumab — Intravitreal bevacizumab (1.5 mg; 0,06 ml) 1 week after baseline; pars plana vitrectomy 3 weeks after baseline
  Other Names: Avastin
  Arms: A
Procedure: pars plana vitrectomy — pars plana vitrectomy 3 weeks after baseline

SUMMARY:
The purpose of this study is to compare the amount of intraoperative intraocular bleeding during 23-gauge pars plana vitrectomy (PPV) for diabetic traction retinal detachment (TRD) with and without preoperative intravitreal bevacizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Macular traction retinal detachment lasting three months or less secondary to diabetic retinopathy.

Exclusion Criteria:

* Massive vitreous hemorrhage preventing from detailed posterior pole examination;
* Previous intra-ocular surgery other than cataract surgery
* Hemodialysis, known bleeding disorders or use of anticoagulants drugs other than aspirin
* Prothrombin time, partial thromboplastin time or platelet count without normal limits
* History of previous thromboembolic events

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
amount of intraoperative intra-ocular bleeding | three weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics Hospital of Ribeirão Preto, School of Medicine of Ribeirão Preto, USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] da R Lucena D, Ribeiro JA, Costa RA, Barbosa JC, Scott IU, de Figueiredo-Pontes LL, Jorge R. Intraoperative bleeding during vitrectomy for diabetic tractional retinal detachment with versus without preoperative intravitreal bevacizumab (IBeTra study). Br J Ophthalmol. 2009 May;93(5):688-91. doi: 10.1136/bjo.2008.151233. Epub 2009 Feb 10. PMID 19208678